CLINICAL TRIAL: NCT06437340
Title: Determinants of Life Satisfaction Levels of Fathers of Children With Cerebral Palsy
Brief Title: Life Satisfaction of Fathers of Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Atahan TURHAN, Dr. Lecturer, Kirsehir Ahi Evran Universitesi
Other Study IDs: KAEU-T.ATAHAN-003
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy; Father-Child Relations; Life Satisfaction
MeSH Terms: conditions — Cerebral Palsy; Personal Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to examine the determinants of life satisfaction among fathers of children diagnosed with Cerebral Palsy.

ELIGIBILITY:
Inclusion Criteria:

* to be literate and to have no communication problems
* to be the father of a child with Cerebral Palsiy (CP) and no other medical diagnosis (aged between 1-18 years)
* to have a child with CP who regularly receives physiotherapy and rehabilitation
* to live in the same house with his wife and child/children
* to be willing to participate in the study

Exclusion Criteria:

* to care for individuals in need of care (such as disabled, elderly, chronically ill) additionally to the child with CP
* to have a chronic disorder (such as neurological, rheumatologic, psychiatric disorder) that would affect life satisfaction.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the Physical Medicine and Rehabilitation Outpatient Clinic with a diagnosis of cerebral palsy were examined by a physiatrist. Children diagnosed with cerebral palsy and their fathers who met the inclusion criteria and agreed to participate in the study were included.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Data | 20week
  Sociodemographic information included gender, age, height, and weight of the children and their fathers. In addition, clinical information about the children, such as duration of physical therapy and type of disability, was recorded.
Satisfaction with Life | 20week
  Life satisfaction level was assessed using the Satisfaction with Life Scale. The scale has a total of 5 items. Participants are asked to rate each item from 1 to 7. The scores obtained from each item can range from 1 to 7, and the total score can range from 1 to 35. The higher the score obtained from the scale, the higher the life satisfaction.
Gross Motor Function | 20week
  The Gross Motor Function Classification System (GMFCS) was used to assess the level of gross motor function in children with Cerebral Palsy (CP). GMFCS is a system that classifies the gross motor function levels of children with CP in the same age groups from 1 to 5. Level 1 represents the highest level of function and level 5 represents the lowest level. A higher level represents a lower level of function.

CONTACTS AND LOCATIONS:
Locations (1):
- Atahan TURHAN, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No